CLINICAL TRIAL: NCT04084522
Title: Effect of Saturated Fat (Desi Ghee) on Gut-Liver Axis in Alcoholic Hepatitis
Acronym: SFAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-SAH-01
Record Dates: First submitted 2019-08-31; First posted 2019-09-10 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-02

CONDITIONS: Alcoholic Hepatitis
Keywords: Alcoholic Hepatitis; Gut Microbiota; Dysbiosis; Malnutrition; Saturated Fat
MeSH Terms: conditions — Hepatitis, Alcoholic; Dysbiosis; Malnutrition | interventions — Ghee

STUDY DESIGN:
Masking Description: As it is a nutritional intervention masking of the either of participants or investigator or other investigator is not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment Group (Placebo Comparator): In addition to standard pharmacological treatment, this group would receive a diet comprising of 35-40 kcal. The total distribution of the calories would be as 55-60% from carbohydrates, 20% from protein and 30% from fat, a fixed amount of 50g of oil would be given and the remaining amount of fat would be met by the invisible dietary fat. The source of visible dietary fat would be refined soyabean oil. This group would not receive any fat in the form of Desi ghee or butter or any nutritional supplement other than the prescribed diet. The diet would be explained to the patient by individual diet charts.
  Interventions: Dietary Supplement: Soyabean Oil
- Intervention Arm (Active Comparator): In addition to standard pharmacological treatment, this group would receive a diet comprising of 35-40kcal and 1.2-1.5gm protein per kg ideal body weight per day. The total distribution of the calories would be as 55-60% from carbohydrates, 20% from protein and 30-35% from fat, a fixed amount of 50g of ghee would be given in 3 divided doses of 30 ml to be taken raw, 20 ml to be used for cooking and the remaining amount of fat would be met by the invisible dietary fat. The source of visible fat would be exclusively Desi ghee. This group would not receive any fat in the form of butter or any other oil or any other nutritional supplement other than the prescribed diet. The diet would be explained to the patient by individual diet charts.
  Interventions: Dietary Supplement: Saturated Fat- Desi Ghee (Clarified Butter)

INTERVENTIONS:
Dietary Supplement: Saturated Fat- Desi Ghee (Clarified Butter) — Desi Ghee which is also known as clarified butter contains around 70% of saturated fat. in India it is one of the important culinary items which promotes longevity and protects against various diseases, attributing numerous health benefits. Ghee consumption has also significant hypolipidemic and hypocholesterolemic effects.
  Arms: Intervention Arm
Dietary Supplement: Soyabean Oil — Soyabean Oil consists of around 84% of unsaturated fat and is the most widely used source of unsaturated fat used in the area.
  Arms: Standard Treatment Group

SUMMARY:
The pathogenesis of the alcoholic liver disease (ALD) is a complex interplay of various etiopathological factors other than direct alcohol toxicity. These factors include inflammation & oxidative stress, dysbiosis, intestinal hyperpermeability, and endotoxemia. Dietary fats not only improve nutritional status in ALD but specific properties of saturated fats (SF) have the potential to favourably modulate these causative factors. This project has two parts, in the animal study 10 groups of murine model of alcoholic hepatitis (AH) would be given SF in the form of Desi Ghee and in the human study patients with AH would be randomized into two groups, one with SF ( Desi Ghee) and the other with usual unsaturated fat (cooking oil). In all effect of SF on gut microbiota, hepatic steatosis, TLR-4 expression, serum adiponectin, endotoxin levels, intestinal tight junction proteins and inflammatory markers in murine models of AH, along with hepatic morbidity & lipid profile, in patients with ALD would be studied.

DETAILED DESCRIPTION:
Alcohol is one of the predominant causes of liver diseases and liver-related deaths worldwide. 10% of heavy drinkers consuming more than 30g /day of alcohol for 5 years develop alcoholic liver disease (ALD). The liver acts as a major organ in alcohol metabolism. Alcohol is metabolized to acetaldehyde, the key toxin in alcohol mediated liver injury which gets converted to reactive oxygen species (ROS) through oxidative pathway thus leading to hepatocyte injury. Several experimental and human studies have shown that alcohol also causes intestinal bacterial overgrowth, intestinal mucosal damage and enhances intestinal permeability, leading to translocation of bacteria and their by-products (like LPS) in the portal circulation. Bacteria further stimulate the production of ROS and pro-inflammatory cytokines like TNF-alpha, IL-6, & chemokines, thus further damaging the liver. Alcohol intake not only causes bacterial overgrowth but also brings a qualitative change in the type of bacteria. The number of gram-negative bacteria like Enterobacteriaceae / Proteobacteria - E.Coli, Firmicutes -Enterococcocus, Bacteriodetes- Fusobacteria and Staphylococaceae -Staphylococcus increase whereas the number of gram-positive bacteria viz. Firmicutes -Lactobacillus, Ruminococcaceae, Lachnospiraceae; Actinobacteria -Bifidobacterium decrease. This change is termed dysbiosis. Thus alcohol-related liver injury is potentiated by alcohol-induced gut barrier dysfunction and ensuing cascade of events, involving dysbiosis. Studies suggest that probiotic administration decreased alcohol-induced dysbiosis, TNF- alpha & IL-6 levels, and improves gut leakiness & liver inflammation. Probiotics also restore the level of lactobacilli thus creating more acidic environment, lowering the intestinal pH & stabilizing mucosal barrier, thereby preventing microbial translocation & blocking TLR-4 signaling cascade and attenuating liver injury. Hence there is evidence that suggests to targeting dysbiosis improves alcohol-related liver disease. Studies have also shown that lactobacilli use saturated fat (SF) for its growth and supplementing SF improves gut lactobacilli levels and subsequently decreases the progression of ALD. Low levels of microbial long-chain saturated fat caused due to alcohol compromise the growth of lactobacillus and hence disrupt gut barrier integrity. A large multicentre epidemiologic study in chronic alcoholics with comparable per capita alcohol intake has shown that intake of saturated fat is associated with lower mortality rates as compared to unsaturated fats (USF) Diet rich in SF has been found to prevent ethanol-induced changes viz. an increase in proteobacteria & liver steatosis, which were actually increased with the consumption of USF. Yet another study reported that the SF diet improved intestinal tight junction expression and alleviated intestinal inflammation caused due to ethanol intake. Supplementation of long-chain fatty SF to ethanol injured mice with increased intestinal permeability restored metabolic homeostasis with decreased intestinal bad bacteria levels where supposedly saturated fat serves as a vitamin B substitute and promotes the growth of lactobacilli species which ameliorates alcoholic liver injury.

Alcohol induced disruption in the intestinal tight junction protein levels, endotoxemia and hepatic LPS signaling were found to be alleviated by SF in the form of medium chain triglycerides. Dietary SF (e.g., palm oil or MCT oil) reversed the established experimental ALD in rats, and improved liver histological changes despite continued intragastric ethanol administration.

Hence the supplementation of SF in ALD is a logical manoeuvre within the nutritional therapy of this disease, as almost 90% of these patients are malnourished primarily due to a reduced diet intake. Fats are concentrated source of energy which makes the food palatable, hence making the attainment of higher calorie (35-40 kcal/kg body weight/day) target possible. With this background use of SF in ALD is a promising modality in the medical armamentarium, given the fact that nutrition remains the cornerstone of the overall therapy.

ELIGIBILITY:
Inclusion Criteria:

All patients with Severe Alcoholic Hepatitis

* Aged between 18-60 years
* Having Maddrey Score of >32
* Last Intake of alcohol from 1 day to 60days
* Patients who agree for complete alcohol abstinence from the day of enrollment

Exclusion Criteria:

Patients with-

* Maddrey Score of <32 and >100
* Comorbidities- Diabetes, Hypertension, Coronary Artery Disease, Chronic Kidney Disease, Hypothyroid
* Continuing Alcohol intake- Non-compliant patients
* Constipation
* On Laxatives until 1 month prior to study
* On probiotics until 1 month prior to study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
To determine the improvement in cirrhosis dysbiosis ratio (CDR) associated with saturated fat in patients with severe alcoholic hepatitis. | 2 months
  The stool sample of the patients would be processed by 16s ribosomal RNA Gene sequencing to observe the diversity, abundance an evenness of the microbial community and thereafter Cirrhosis dysbiosis ratio (CDR) would be calculated at the starting and the end of the study i.e at baseline and at the end of two months.

SECONDARY OUTCOMES:
To study the serum endotoxin (lipoploysacchride) levels in patients with severe alcoholic hepatitis | 2 months
  The collected blood sample would be assessed for endotoxin levels by using Toxin Sensor TM Chromogenic LAL Endotoxin Assay Kit

OTHER OUTCOMES:
To study the serum pro- inflammatory marker, TNF-alpha in patients with severe alcoholic hepatitis | 2 months
  The collected blood sample would be assessed for TNF- alpha levels by using Quantikine ELISA kit
To study the serum pro- inflammatory marker, IL-6 in patients with severe alcoholic hepatitis | 2 months
  The collected blood sample would be assessed for IL-6 levels by using Quantikine ELISA kit
To study the serum pro- inflammatory marker, NF-kB in patients with severe alcoholic hepatitis | 2 months
  The collected blood sample would be assessed for NF-kB levels by using Quantikine ELISA kit
To study the serum anti- inflammatory marker,adiponectin in patients with severe alcoholic hepatitis | 2 months
  The collected blood sample would be assessed for adiponectin levels by using Quantikine ELISA kit
To study the serum anti- inflammatory marker, IL-10 in patients with severe alcoholic hepatitis | 2 months
  The collected blood sample would be assessed for IL-10 levels by using Quantikine ELISA kit
To observe the expression of gut microbiome specific genes in patients with severe alcoholic hepatitis | 2 months
  The stool sample collected would be assessed for Fab genes (G and F) expression using 16s ribosomal gene sequencing.
To observe Clinical benefit in patients of severe alcoholic hepatitis | 2 months
  Clinical benefit in terms of resolution of signs & symptoms to be observed.
To observe Clinical benefit in patients of severe alcoholic hepatitis | 2 months
  Clinical benefit in terms of improvement in Bilirubin levels to be observed
To observe Clinical benefit in patients of severe alcoholic hepatitis | 2 months
  Clinical benefit in terms of reduction of AST & ALT levels to be observed
To observe Clinical benefit in patients of severe alcoholic hepatitis | 2 months
  Clinical benefit in terms of reduction Maddrey Score to be observed
To observe the Nutritional status in patients with Severe Alcoholic hepatitis | 2 months
  Body composition analysis by BIA (Bioelectrical impedance analysis) for nutritional screening of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jaya Benjamin, PhD, Principal Investigator — Associate Professor
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edenberg HJ. The genetics of alcohol metabolism: role of alcohol dehydrogenase and aldehyde dehydrogenase variants. Alcohol Res Health. 2007;30(1):5-13. PMID 17718394
- [Background] Keshavarzian A, Farhadi A, Forsyth CB, Rangan J, Jakate S, Shaikh M, Banan A, Fields JZ. Evidence that chronic alcohol exposure promotes intestinal oxidative stress, intestinal hyperpermeability and endotoxemia prior to development of alcoholic steatohepatitis in rats. J Hepatol. 2009 Mar;50(3):538-47. doi: 10.1016/j.jhep.2008.10.028. Epub 2008 Dec 29. PMID 19155080
- [Background] Mutlu E, Keshavarzian A, Engen P, Forsyth CB, Sikaroodi M, Gillevet P. Intestinal dysbiosis: a possible mechanism of alcohol-induced endotoxemia and alcoholic steatohepatitis in rats. Alcohol Clin Exp Res. 2009 Oct;33(10):1836-46. doi: 10.1111/j.1530-0277.2009.01022.x. Epub 2009 Jul 23. PMID 19645728
- [Background] Su GL, Rahemtulla A, Thomas P, Klein RD, Wang SC, Nanji AA. CD14 and lipopolysaccharide binding protein expression in a rat model of alcoholic liver disease. Am J Pathol. 1998 Mar;152(3):841-9. PMID 9502426
- [Background] Hritz I, Mandrekar P, Velayudham A, Catalano D, Dolganiuc A, Kodys K, Kurt-Jones E, Szabo G. The critical role of toll-like receptor (TLR) 4 in alcoholic liver disease is independent of the common TLR adapter MyD88. Hepatology. 2008 Oct;48(4):1224-31. doi: 10.1002/hep.22470. PMID 18792393
- [Background] Nanji AA, Jokelainen K, Tipoe GL, Rahemtulla A, Dannenberg AJ. Dietary saturated fatty acids reverse inflammatory and fibrotic changes in rat liver despite continued ethanol administration. J Pharmacol Exp Ther. 2001 Nov;299(2):638-44. PMID 11602676
- [Background] Kirpich IA, Petrosino J, Ajami N, Feng W, Wang Y, Liu Y, Beier JI, Barve SS, Yin X, Wei X, Zhang X, McClain CJ. Saturated and Unsaturated Dietary Fats Differentially Modulate Ethanol-Induced Changes in Gut Microbiome and Metabolome in a Mouse Model of Alcoholic Liver Disease. Am J Pathol. 2016 Apr;186(4):765-76. doi: 10.1016/j.ajpath.2015.11.017. PMID 27012191
- [Background] Kirpich IA, Solovieva NV, Leikhter SN, Shidakova NA, Lebedeva OV, Sidorov PI, Bazhukova TA, Soloviev AG, Barve SS, McClain CJ, Cave M. Probiotics restore bowel flora and improve liver enzymes in human alcohol-induced liver injury: a pilot study. Alcohol. 2008 Dec;42(8):675-82. doi: 10.1016/j.alcohol.2008.08.006. PMID 19038698
- [Background] Chen P, Torralba M, Tan J, Embree M, Zengler K, Starkel P, van Pijkeren JP, DePew J, Loomba R, Ho SB, Bajaj JS, Mutlu EA, Keshavarzian A, Tsukamoto H, Nelson KE, Fouts DE, Schnabl B. Supplementation of saturated long-chain fatty acids maintains intestinal eubiosis and reduces ethanol-induced liver injury in mice. Gastroenterology. 2015 Jan;148(1):203-214.e16. doi: 10.1053/j.gastro.2014.09.014. Epub 2014 Sep 16. PMID 25239591
- [Background] Kirpich IA, Feng W, Wang Y, Liu Y, Barker DF, Barve SS, McClain CJ. The type of dietary fat modulates intestinal tight junction integrity, gut permeability, and hepatic toll-like receptor expression in a mouse model of alcoholic liver disease. Alcohol Clin Exp Res. 2012 May;36(5):835-46. doi: 10.1111/j.1530-0277.2011.01673.x. Epub 2011 Dec 7. PMID 22150547
- [Background] Zhong W, Li Q, Xie G, Sun X, Tan X, Sun X, Jia W, Zhou Z. Dietary fat sources differentially modulate intestinal barrier and hepatic inflammation in alcohol-induced liver injury in rats. Am J Physiol Gastrointest Liver Physiol. 2013 Dec;305(12):G919-32. doi: 10.1152/ajpgi.00226.2013. Epub 2013 Oct 10. PMID 24113767
- See also: Pubmed has been used for all the papers search. — https://www.ncbi.nlm.nih.gov/pubmed/